CLINICAL TRIAL: NCT01512420
Title: A Multicenter, Prospective, Observational Study to Identify Different Prognostic Factors Related to Survival in Patients With Previously Treated Advanced NSCLC With Wild-type Epidermal Growth Factor Receptor (EGFR) Gene.
Brief Title: An Observational Study of Tarceva (Erlotinib) in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer With Wild-Type Epidermal Growth Factor Receptor (EGFR) Gene (WILT)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27773
Record Dates: First submitted 2011-12-19; First posted 2012-01-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of second-line Tarceva (erlotinib) in patients with previously treated advanced non-small cell lung cancer with confirmed wild-type epidermal growth factor receptor (EGFR) gene. The aim of the study is to identify from baseline clinical and demographic patient characteristics prognostic factors related to overall survival with second-line Tarceva treatment. Data will be collected from eligible patients for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC)
* Patients with known wild-type EGFR gene; patients with unknown EGFR mutation status are allowed if they fulfil the following criteria:
* squamous cell carcinoma lung cancer histology, and
* current smoker, or former smoker who has stopped smoking less than 10 years ago and has had a total of >15 pack-years of smoking
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Patients having failed one prior chemotherapy regimen and eligible for a second-line treatment with Tarceva

Exclusion Criteria:

* Current treatment with an investigational drug or participation in another investigational study
* Severe or uncontrolled systemic disease, active infection, concomitant malignancy or a second primary malignancy except for in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin
* Clinically active interstitial lung disease
* Recent myocardial infarction or unstable angina
* Progressive or uncontrolled brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously treated advanced NSCLC, with wild-type EGFR gene or squamous cell carcinoma histology
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Correlation of overall survival with baseline clinical/demographic patient characteristics | approximately 2 years
Correlation of overall survival with baseline tumour characteristics | approximately 2 years
Correlation of overall survival with previous treatment regimens | approximately 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR), tumour assessments according to RECIST criteria | approximately 2 years
Disease control rate | approximately 2 years
Progression-free survival | approximately 2 years
Safety: Incidence of adverse events | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- Spain (32):
  - Vitoria-Gasteiz, Alava
  - Elda, Alicante
  - Maó, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Cáceres, Caceres
  - Santander, Cantabria
  - Girona, Girona
  - Donostia / San Sebastian, Guipuzcoa
  - Barbastro, Huesca
  - Huesca, Huesca
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Logroño, La Rioja
  - Las Palmas de Gran Canaria, Las Palmas
  - León, Leon
  - Lugo, Lugo
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - Melilla, Malaga
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
  - Reus, Tarragona
  - San Cristóbal de La Laguna, Tenerife
  - Teruel, Teruel
  - Toledo, Toledo
  - Valencia, Valencia
  - Xàtiva, Valencia
  - Valladolid, Valladolid
  - Bilbao, Vizcaya
  - Zamora, Zamora
  - Zaragoza, Zaragoza